CLINICAL TRIAL: NCT05839301
Title: A Single-center, Randomized, Double-blind Trial to Evaluate the Lot-to-lot Consistency of Live Attenuated Varicella Vaccine in Healthy People 1-12 Years of Age
Brief Title: A Trial to Evaluate the Lot-to-lot Consistency of Live Attenuated Varicella Vaccine in Healthy People 1-12 Years of Age
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry); Jiangsu Province Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CNBG-BIBP-VZV-08
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Varicella
Keywords: varicella vaccine; safety; immunogenicity; lot-to-lot consistency
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Group1 (Experimental): Single subcutaneous injection of the investigational vaccine (0.5ml)
  Interventions: Biological: Investigational live attenuated varicella vaccine (lot 1)
- Experimental Group2 (Experimental): Single subcutaneous injection of the investigational vaccine (0.5ml)
  Interventions: Biological: Investigational live attenuated varicella vaccine (lot 2)
- Experimental Group3 (Experimental): Single subcutaneous injection of the investigational vaccine (0.5ml)
  Interventions: Biological: Investigational live attenuated varicella vaccine (lot 3)

INTERVENTIONS:
Biological: Investigational live attenuated varicella vaccine (lot 1) — 0.5ml/vial
  Arms: Experimental Group1
Biological: Investigational live attenuated varicella vaccine (lot 2) — 0.5ml/vial
  Arms: Experimental Group2
Biological: Investigational live attenuated varicella vaccine (lot 3) — 0.5ml/vial
  Arms: Experimental Group3

SUMMARY:
The goal of this clinical trial is to evaluate the lot-to-lot consistency, immunogenicity, and safety of live attenuated varicella vaccine manufactured by Beijing Institute of Biological Products Co., Ltd in healthy children.

DETAILED DESCRIPTION:
This trial is aim to evaluate the lot-to-lot consistency, immunogenicity, and safety of live attenuated varicella vaccine manufactured by Beijing Institute of Biological Products Co., Ltd in healthy people 1 to 12 years of age.1200 healthy subjects aged 1-12 years were enrolled after their guardians passed the informed consent, inclusion and exclusion criteria screening in turn. Three batches were randomized in a 1:1: 1 ratio, with 400 subjects in each batch.All subjects received 1 dose of trial vaccine (Batch 1 or Batch 2 or Batch 3) and all were collected Blood samples were collected from subjects before vaccination, on Day 30 after vaccination for serum neutralizing antibody testing to evaluate immunogenicity, and Safety observations were performed until 6 months post-vaccination in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to 12 years on the day of enrollment ,male or female, and able to provide legal identity certificate.
* Subjects and/or guardians have the ability to understand the study requirements and process, agree to participate in the clinical trial and sign the informed consent form.
* Axillary temperature ≤ 37.0 ° C on the day of enrollment.

Exclusion Criteria:

* Previous vaccination against varicella (eg, varicella vaccine, measles + varicella vaccine).
* History of varicella or herpes zoster infection, or exposure to varicella/herpes zoster within 30 days of enrollment or suspected varicella/herpes zoster;
* Current use of salicylates (including salicylic acid, aspirin, diflunisal, p-aminosalicylic acid (sodium), salsalsalate, benorilate, etc.), or planned long-term use during the study.
* Febrile illness (axillary temperature ≥ 38.5 ° C) or use of antipyretic, analgesic, and anti-allergic drugs (eg, acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) 3 days before vaccination.
* History of allergy to vaccine ingredients and excipients or severe drug allergy, such as anaphylactic shock, allergic laryngeal edema, Henoch-Schonlein purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), severe urticaria.
* History of epilepsy, convulsions, or convulsions, or a family history of psychosis.
* Impaired immune function or has been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune diseases.
* Patients suffering from serious congenital malformations, genetic diseases, serious cardiovascular diseases, serious liver/kidney diseases, diabetes with complications, malignant tumors, severe malnutrition.
* Immunosuppressant therapy such as chronic oral or injectable glucocorticoid therapy (≥ 14 days at doses ≥ 2 mg/kg/day or ≥ 20 mg/day prednisone or equivalent prednisone dose) within 3 months prior to administration of trial vaccine or planned 30 days following administration, but not limited by topical use (eg, ointment, eye drops, inhalers, or nasal sprays).
* Receiving blood/blood-related products or immunoglobulins 3 months before vaccination or planning to use such products 30 days after vaccination.
* Vaccination with a live attenuated vaccine within 30 days or any vaccine within 14 days prior to vaccination.
* Absence of spleen or splenectomy due to any condition such as splenectomy.
* Patients with a history of thrombocytopenia or other coagulation disorders, which may cause contraindications to subcutaneous injection.
* Infectious, suppurative and allergic skin diseases.
* Participating in other investigational or non-registered product (drug, vaccine or device, etc.) clinical trials, or planning to participate in other clinical trials before the end of this clinical trial.
* Subject has any other factor that, in the judgment of the investigator, would make the subject unsuitable for participation in the clinical trial.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titers (GMT) of anti-VZV neutralizing antibodies | 30 days after vaccination
  Geometric mean titers (GMT) of anti-VZV neutralizing antibodies 30 days after vaccination in the negative population before immunization

SECONDARY OUTCOMES:
Positive conversion rate and geometric mean fold increase (GMFI) of anti-VZV neutralizing antibodies | 30 days after vaccination
  Positive conversion rate and geometric mean fold increase (GMFI) of anti-VZV neutralizing antibodies 30 days after vaccination in the negative population before immunization
Positive conversion rate, GMT, and GMFI of anti-VZV neutralizing antibodies | 30 days after vaccination
  Positive conversion rate, GMT, and GMFI of anti-VZV neutralizing antibodies 30 days after vaccination in the whole population
The incidences of adverse events (AEs) | 30 days after vaccination
  AEs occurred witnin 30 days after vaccination will be collected
The incidences of serious adverse events (SAEs) and Adverse Event of Special Interest(AESI) | 6 months after vaccination
  SAEs and AESI occurred witnin 6 months after vaccination will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Principal Investigator — Jiangsu Province Centers for Disease Control and Prevention
Locations (1):
- Xinyi Center for Disease Control and Prevention, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No